CLINICAL TRIAL: NCT07284875
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of KAI-9531 Administered Once Weekly in Participants Living With Obesity or Overweight With Weight-Related Comorbidities Who Do Not Have Diabetes
Brief Title: Efficacy and Safety of KAI-9531 in Participants Living With Obesity or Overweight With Weight-Related Comorbidities Who Do Not Have Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kailera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K9531-3103; 2025-523486-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: Overweight; Obesity; KAI-9531; Glucagon-like Peptide-1; GLP-1; Glucose-dependent Insulinotropic Peptide; GIP
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- KAI-9531: Dose 1 (Experimental): Participants will receive Dose 1 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- KAI-9531: Dose 2 (Experimental): Participants will receive Dose 2 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- KAI-9531: Dose 3 (Experimental): Participants will receive Dose 3 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- KAI-9531: Dose 4 (Experimental): Participants will receive Dose 4 of KAI-9531 once weekly.
  Interventions: Drug: KAI-9531
- Placebo (Placebo Comparator): Participants will receive placebo matched to KAI-9531 once weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAI-9531 — SC Injection
  Arms: KAI-9531: Dose 1; KAI-9531: Dose 2; KAI-9531: Dose 3; KAI-9531: Dose 4
Drug: Placebo — SC Injection
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the effects of KAI-9531 subcutaneous (SC) injection once weekly compared to placebo on percent change in body weight.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m^2 or BMI ≥27 kg/m^2 and previously diagnosed with at least 1 of the following:

  1. hypertension,
  2. dyslipidemia,
  3. obstructive sleep apnea, or
  4. cardiovascular (CV) disease.
* History of at least 1 self-reported unsuccessful effort to lose weight with diet and exercise within the prior 6 months.

Exclusion Criteria:

* Current diagnosis or history of diabetes mellitus.
* Started medications within 3 months prior to Screening that may cause significant weight gain, including, but not limited to, tricyclic antidepressants, atypical antipsychotics, and mood stabilizers.
* Unstable weight defined as self-reported change in body weight exceeding 5% within 3 months prior to Screening.
* Family or personal history of multiple endocrine neoplasia Type 2 or medullary thyroid cancer.
* Uncontrolled hypertension or unstable cardiovascular disease.
* History of chronic or acute pancreatitis.
* Known clinically significant gastric-emptying abnormality or chronic treatment with medications that directly affect gastrointestinal motility.
* History of suicide attempt.
* History of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder.
* Received treatment with semaglutide, tirzepatide, GLP-1 receptor agonist, GLP-1/glucose-dependent insulinotropic polypeptide (GIP), or glucagon receptor agonist within 3 months prior to Screening.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
Dose 3 and 4 versus Placebo: Percent Change From Baseline in Body Weight at Week 76 | Baseline, Week 76

SECONDARY OUTCOMES:
Dose 1 and 2 versus Placebo: Percent Change From Baseline in Body Weight at Week 76 | Baseline, Week 76
Percentage of Participants with ≥5%, ≥10%, ≥15%, ≥20% and ≥25% Reduction in Body Weight | Baseline, Week 76
Change From Baseline in Waist Circumference | Baseline, Week 76
Change From Baseline in Absolute Body Weight | Baseline, Week 76
Change From Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 76
Percent Change From Baseline in Fasting Triglycerides | Baseline, Week 76
Percent Change From Baseline in Fasting High-density Lipoprotein (HDL)-cholesterol | Baseline, Week 76
Percent Change From Baseline in Fasting Non-HDL-cholesterol | Baseline, Week 76
Change From Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score | Baseline, Week 76
Participants with Body Mass Index (BMI) ≥35 Kilograms per Square Meter (kg/m^2): Percent Change From Baseline in Body Weight | Baseline, Week 76
Percentage of Participants with ≥30% Reduction in Body Weight | Baseline, Week 76
Change From Baseline in BMI | Baseline, Week 76
Change From Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 76
Percent Change From Baseline in Total Cholesterol | Baseline, Week 76
Percent Change From Baseline in Low-density Lipoprotein (LDL)-cholesterol | Baseline, Week 76
Percent Change From Baseline in Very Low-density Lipoprotein (VLDL)-cholesterol | Baseline, Week 76
Percent Change From Baseline in Fasting Insulin | Baseline, Week 76
Change From Baseline in Fasting Blood Glucose | Baseline, Week 76
Change From Baseline in Control of Eating Questionnaire (CoEQ) Craving Control Score | Baseline, Week 76
Change From Baseline in CoEQ Positive Mood Score | Baseline, Week 76
Change From Baseline in CoEQ Craving for Sweets Score | Baseline, Week 76
Change From Baseline in CoEQ Craving for Savory Food Score | Baseline, Week 76
Change From Baseline in CoEQ Hunger Score | Baseline, Week 76
Change From Baseline in CoEQ Satiety Score | Baseline, Week 76
Change From Baseline in CoEQ Combined Score | Baseline, Week 76
Change From Baseline in Food Noise Questionnaire (FNQ) Score | Baseline, Week 76
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Week 80
Number of Participants With Anti-drug Antibodies (ADAs) | Up to Week 80
Number of Participants With Neutralizing Antibodies (Nabs) | Up to Week 80
Plasma Concentrations of KAI-9531 | Up to Week 76

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Kailera Clinical Site, Anniston, Alabama
  - Kailera Clinical Site, Aurora, Colorado
  - Kailera Clinical Site, Bridgeport, Connecticut
  - Kailera Clinical Site, Columbia, Maryland
  - Kailera Clinical Site, Rochester, New York
  - Kailera Clinical Site, Morehead City, North Carolina
  - Kailera Clinical Site, Chickasha, Oklahoma
  - Kailera Clinical Site, Chattanooga, Tennessee
  - Kailera Clinical Site, Amarillo, Texas
  - Kailera Clinical Site, DeSoto, Texas
  - Kailera Clinical Site, Tomball, Texas
  - Kailera Clinical Site, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No